CLINICAL TRIAL: NCT06695858
Title: The Incidence of Post-Operative Lung Atelectasis With Erector Spinae Plane Block in Bariatric Surgery: A Prospective Randomized Controlled Trial
Brief Title: The Incidence of Post-Operative Lung Atelectasis With Erector Spinae Plane Block in Bariatric Surgery:
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MD-271-2023
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Atelectasis; Bariatric Surgery
Keywords: Ultrasound; Erector spinae; Bariatric surgery; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: An experienced anesthetist will open the envelopes, prepare the local anesthetics, and perform the assigned technique with no further involvement in the study.
  A blinded investigator (an anesthesia and pain therapy specialist) will be responsible for perioperative data collection, pain assessment during the first 24 postoperative hours, and providing analgesia. All patients were blinded to the assigned technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): Patients received bilateral sham ultrasound-guided ESPB using 20 mL normal saline on each side.
  Interventions: Drug: ESPB
- ESPB group (Experimental): Patients received bilateral ultrasound-guided ESPB using 20 mL bupivacaine 0.25% on each side.
  Interventions: Drug: ESPB

INTERVENTIONS:
Drug: ESPB — Patients received bilateral ultrasound-guided ESPB using 20 mL bupivacaine 0.25% on each side.

SUMMARY:
We aim to compare the incidence of post-operative lung atelectasis with erector spinae plane block versus systemic analgesia in patients undergoing bariatric surgery

DETAILED DESCRIPTION:
Patients will be randomly allocated at a 1:1 ratio into two groups, using a computer-generated random sequence and concealed envelopes that contained group assignments and drug preparation instructions.

Group I (control group): Patients received bilateral sham ultrasound-guided ESPB using 20 mL normal saline on each side.

Group II (ESPB group): Patients received bilateral ultrasound-guided ESPB using 20 mL bupivacaine 0.25% on each side.

An experienced anesthetist will open the envelopes, prepare the local anesthetics, and perform the assigned technique with no further involvement in the study.

A blinded investigator (an anesthesia and pain therapy specialist) will be responsible for perioperative data collection, pain assessment during the first 24 postoperative hours, and providing analgesia. All patients were blinded to the assigned technique.

Upon arrival to the operating room, routine monitors (ECG, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and prophylactic antiemetic will be provided in the form of slow intravenous injection of 8 mg dexamethasone drugs. The study protocol, the numeric rating scale (NRS) of pain, and the use of patient-controlled analgesia (PCA) device will be explained to each participant during the preoperative anesthesia counseling.

Then patients will receive either ultrasound-guided bilateral ESPB or sham block according to their group allocation.

The severity of atelectasis will be evaluated by calculating the modified lung ultrasound score from Monastesse et al. [15], with scores between 0 and 3 (0=≤2 B lines; 1=≥3 B lines or multiple areas of subpleural consolidation separated by a normal pleural line; 2=multiple coalescent B lines, or multiple areas of subpleural consolidation separated by a thickened pleura; 3=consolidation or small areas of subpleural consolidation >1×2 cm in diameter (Supplementary Table 1). Lung ultrasound score 0 to 36 was estimated by summing the 12 individual quadrant scores. pulmonary atelectasis will be defined to be significant when the lung ultrasound score ≥2 in any region. We assumed that the lung ultrasound score on T4 can reflect the primary outcomes.

Anesthesia Dexamethasone (4mg to 8mg) will be given one hour before operation as a prophylaxis from nusea and vomiting.

Anesthesia will be induced with 2 mg/kg propofol, 2 mcg/kg fentanyl (lean body weight), and tracheal intubation will be facilitated by 0.6 mg/kg ideal body weight rocuronium after loss of consciousness. Anesthesia will be maintained with isoflurane 1-1.2% in oxygen and 0.1 mg/kg rocuronium every 30 minutes. Arterial catheter will be inserted for blood sampling and invasive blood pressure monitoring.

Fluid management Intraoperative fluid management included a baseline infusion of crystalloids at the rate of 4 mL/kg/h and further fluid administration will be according to the attending anesthetist discretion aided by the pulse pressure variation in accordance with the local protocols of our hospital [16].

Ventilation All patients will receive volume control ventilation with tidal volume of 6-8 mL/kg of predicted body weight, positive end expiratory pressure (PEEP) of 5 cm H2O, fraction of inspired oxygen (FiO2) of 40%, and respiratory rate will be adjusted to maintain end-tidal CO2 of 30-40 mmHg. Surgery will be performed in reverse Trendelenburg position 30-40 degrees and the pneumoperitoneum will be standardized with an abdominal pressure at 12 cm H2O.

Intraoperative inadequate analgesia, indicated by increase of the heart rate (HR) or the mean arterial blood pressure (MAP) more than 20% above the baseline, will be managed using fentanyl 1 μg/kg. Intraoperative fentanyl consumption will be calculated.

Prevention of postoperative nausea and vomiting will be attempted using 4 mg ondansetron at the end of surgery. IV paracetamol 1g and ketorolac 30 mg will be administered to all patients 10 minutes before the end of surgery. At the end of surgery, muscle relaxant will be reversed using neostigmine 0.05 mg/kg and atropine 0.02 mg/kg. Awake extubation will be established after adequate reversal of neuromuscular block.

Patients will be transported to the post-anesthesia care unit (PACU). In the PACU, patients will be placed in the semi-sitting position, Postoperative pain will be assessed using NRS (where 0 corresponds to no pain and 10 to the worst pain) at PACU admission and 30 minutes, 1, 2, 4, 6, 8, 12, 18, and 24 hours postoperatively.

Criteria for intensive care unit (ICU) admission will be either respiratory-related, such as shortness of breath or desaturation (SpO2 < 90%), or non-respiratory-related, such as anastomotic leak or bleeding.

In PACU, bolus dose of morphine; 50mcg/kg will be given by the physician if pain score of the patient is more than 4. All patients with NRS ≤ 4 will receive morphine via an infusion pump (Zhejiang Fert disposable infusion pump 275ml with constant flow 5ml/hour. Zhejiang Fert Medical Device Co.,Ltd). Patients will receive a morphine continuous infusion of 10mcg/kg/hour (maximum 1 mg/hour). The patients will be instructed to report any pain to a pain nurse, and if the NRS increase to more than 4, the pain nurse will inform the anaesthesiologist. Inadequate analgesia (NRS more than 4) will be treated with a clinician bolus of 50mcg/kg with a time interval of 30 minutes at least between the additional doses till NRS decreases to less than 4 [17]. If the patient appeared sedated (Ramsay sedation scale > 2) [18].and/or severe morphine-related side effects are encountered including respiratory depression (Spo2 < 95% and/or respiratory rate < 12 breaths/min), allergic reaction, hypotension, or severe pruritus, will be treated by stopping the pump until appropriate recovery and by a decrease in the demand dose of 20%.

Any intraoperative or postoperative complications were recorded. In case of vomiting, metoclopramide 10 mg will be given. Ondansetron 8mg will be given in persistent vomiting. In case of respiratory depression, Naloxone 1mcg/kg will be administered and oxygen will be supplied by oxygen mask. In case of decrease in MABP>20% from base line, the patient will receive a 500 ml ringer infusion with 5 mg ephedrine. If HR decrease to 45 beats/minute, atropine 0.5 mg will be given.

ELIGIBILITY:
Inclusion Criteria:

* patients with body mass index ≥35 kg/m2
* scheduled to undergo laparoscopic bariatric surgery.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical class> III.
* Subjects with contraindications to peripheral regional anesthesia blocks
* neurological or psychological disorders
* inability to cooperate
* pre-existing chronic pain or cognitive dysfunction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-10-18 (Actual); Study Completion 2025-10-18 (Actual)

PRIMARY OUTCOMES:
Lung atelectasis | 6 hours
  Lung atelectasis (defined as lung ultrasound score ≥2 in any lung region)

SECONDARY OUTCOMES:
NRS | 24 hours
  pain will be assessed using numerical rating score

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided